CLINICAL TRIAL: NCT02070796
Title: Single-site, Open-label, Randomized, Cross-over Study in Healthy Chinese Subjects to Evaluate the Bioequivalence of Single-dose Rotigotine Transdermal Patch (2 mg/24 h) Comparing 2 Different Formulations
Brief Title: Single-site, Open-label, Randomized, Cross-over Study in Healthy Chinese Subjects to Evaluate the Bioequivalence of Single-dose Rotigotine Transdermal Patch Comparing 2 Different Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PD0011
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Rotigotine; Transdermal Patch; Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment A - B (Experimental): Single application of the test transdermal patch (Treatment A, Rotigotine PR2.2.1) for 24 hours, followed by a Wash-Out Period of 7 days and a single application of the reference transdermal patch (Treatment B, Rotigotine PR2.1.1) for 24 hours.
  Interventions: Drug: Rotigotine PR2.2.1; Drug: Rotigotine PR2.1.1
- Treatment B - A (Active Comparator): Single application of the reference transdermal patch (Treatment B, Rotigotine PR2.1.1) for 24 hours, followed by a Wash-Out Period of 7 days and a single application of the test transdermal patch (Treatment A, Rotigotine PR2.2.1) for 24 hours.
  Interventions: Drug: Rotigotine PR2.2.1; Drug: Rotigotine PR2.1.1

INTERVENTIONS:
Drug: Rotigotine PR2.2.1 — Treatment A:
  Rotigotine Transdermal patch 2 mg/24 hr (10 cm^2) Test drug product PR2.2.1. Single application of 1 patch for 24 hours.
Drug: Rotigotine PR2.1.1 — Treatment B:
  Rotigotine Transdermal patch 2 mg/24 hr (10 cm^2) Reference drug product PR2.1.1. Single application of 1 patch for 24 hours.

SUMMARY:
The primary objective of the study is to establish Bioequivalence (BE) of 2 different formulations of the 2 mg/24 hr (10 cm^2) Rotigotine transdermal patches in Chinese subjects.

DETAILED DESCRIPTION:
Bioequivalence will be concluded if the 90 % Confidence Intervals (CIs) for the ratio Treatment A/Treatment B are fully included in the acceptance range from 0.8-1.25 for AUC(0-t) and AUC, and within the acceptance range from 0.7 to 1.43 for Cmax.

ELIGIBILITY:
Inclusion Criteria:

* An Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject
* Subject is considered reliable and capable of adhering to the protocol, visit schedule, and patch application according to the judgment of the investigator
* Subject is willing and able to comply with all study requirements
* Subject is Chinese (with all 4 grandparents being of Chinese origin, as well), male, and aged between 18 and 40 years (inclusive)
* Subject is healthy (no clinically significant findings in any of the investigations at the Eligibility Assessment (EA))
* Subject has a body mass index between 19 kg/m² and 24 kg/m² (inclusive), and a body weight greater than or equal to 50 kg
* Subject agreed to practice a medically accepted method of contraception (eg, condom, spermicide) unless sexually abstinent for the duration of the study and up to 3 months after the final patch application

Exclusion Criteria:

* Subject has previously participated in this study or subject has previously been assigned to treatment in a Rotigotine study
* Subject has participated in another study of an Investigational Medicinal Product (IMP) (or a medical device) within the previous 3 months or is currently participating in another study of an IMP (or a medical device)
* Subject has a history of diagnosis, counseling, or treatment for chronic alcohol or drug abuse within the previous 2 years
* Subject has a known clinically significant allergy or known or suspected clinically significant drug hypersensitivity to any components of the IMP or comparable drugs that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject has lifetime history of suicide attempt
* Subject has a history of significant skin hypersensitivity to adhesives or other transdermal products or has recently unresolved contact dermatitis
* Subject has an medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject has a history or present condition of epilepsy and/or seizures
* Subject has a history or present condition of an atopic or eczematous dermatitis, psoriasis, and/or an active skin disease

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration (AUC(0-t)) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application.
Area under the plasma concentration-time curve from zero up to Infinity (AUC) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
The maximum plasma concentration of unconjugated Rotigotine (Cmax) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by apparent dose (mg) (AUC(0-t) norm (apparent dose)) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by body weight (kg) (AUC(0-t) norm (BW)) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Area under the plasma concentration-time curve from zero up to infinity normalized by apparent dose (mg) (AUCnorm (apparent dose)) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Area under the plasma concentration-time curve from zero up to infinity normalized by body weight (kg) (AUCnorm (BW)) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Maximum plasma concentration of unconjugated Rotigotine normalized by apparent dose (Cmax, norm (apparent dose)) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Maximum plasma concentration of unconjugated Rotigotine normalized by body weight (Cmax, norm (BW)) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Time to reach a maximum plasma concentration of unconjugated Rotigotine after patch application (tmax) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Mean residence time (MRT) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Rate constant of elimination (λz) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Terminal half-life (t1/2) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Relative bioavailability calculated based on Cmax (fCmax) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Relative bioavailability calculated based on AUC (fAUC) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application
Apparent total body clearance (CL/f) | Blood samples will be taken predose, and at 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 16 hr, 24 hr (immediately prior to patch removal in the morning of Day 2), 25 hr, 26 hr, 28 hr, 30 hr, 32 hr, 36 hr, 40 hr, and 48 hr after patch application

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Hong Kong, China

REFERENCES:
- [Derived] Liu Y, Tomlinson B, Guo J, Asgharnejad M, Bauer L, Surmann E, Guo X, Elshoff JP. Pharmacokinetics, Tolerability, and Bioequivalence of Two Formulations of Rotigotine in Healthy Chinese Subjects. Clin Ther. 2018 Jul;40(7):1108-1121.e8. doi: 10.1016/j.clinthera.2018.05.009. PMID 30098648